CLINICAL TRIAL: NCT01869049
Title: A Study on the Alteration of Macrophage Function in the Spleen Tissue From Patients With Primary Immune Thrombocytopenia (ITP): a Multicenter, Perspective, Clinical Trial
Brief Title: The Alteration of Macrophage Function in the Spleen Tissues From Patients With Primary Immune Thrombocytopenia
Acronym: ITP
Status: Withdrawn | Type: Observational
Why Stopped: No eligible patient was enrolled.
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Ming Hou, professor, Shandong University
Other Study IDs: ITP-Spleen; 81070396 (Other Grant/Funding Number: Natural Science Foundation of China)
Record Dates: First submitted 2013-04-03; First posted 2013-06-05 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2013-04

CONDITIONS: Immune Thrombocytopenia
Keywords: Immune Thrombocytopenia; macrophage; spleen tissue
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The biospecimens were retained for PCR, western blotting and FACS analysis.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ITP patients accepted splenectomy
- Trauma with spleen rupture underwent splenectomy

SUMMARY:
This project was undertaken by Qilu Hospital of Shandong University and other well-known hospitals in China. In order to report the alteration on the macrophage function in the spleen tissue of primary immune thrombocytopenia (ITP).

ELIGIBILITY:
Inclusion Criteria:

* adult ITP patients whose platelet counts remain less than 10 x 10^9/L
* patients whose platelet counts remain less than 30 x 10^9/L and who continue to experience excessive bleeding after 4 to 6 weeks of appropriate medical treatment
* patients who have experienced a transient response to primary treatment and have platelet counts less than 30 x 10^9/L after 3 months
* require continuous glucocorticoid therapy to maintain safe platelet counts
* Willing and able to sign written informed consent.

Exclusion Criteria:

* Received chemotherapy or anticoagulants or other drugs affecting the platelet counts within 3 months before the screening visit.
* Current HIV infection or hepatitis B virus or hepatitis C virus infections.
* Severe medical condition (lung, hepatic or renal disorder) other than chronic ITP. Unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure, uncontrolled hypertension or cardiac arrhythmia)
* Female patients who are pregnant.
* Have a known diagnosis of other autoimmune diseases, established in the medical history and laboratory findings with positive results for the determination of antinuclear antibodies, anti-cardiolipin antibodies, lupus anticoagulant or direct Coombs test.
* Patients who are deemed unsuitable for the study by the investigator.

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chinese Adult with primary immune thrombocytopenia
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation of platelet response (Complete Response) | The time frame is up to 3 months per subject
  CR. A complete response (CR) was defined as a sustained (≥ 3 months) platelet count ≥ 100×10^9/L without recurrence of thrombocytopenia
Evaluation of platelet response (R) | The time frame is up to 3 months per subject
  R. A response (R) was defined as a sustained (≥ 3 months) platelet count ≥ 30×10^9/L without recurrence of thrombocytopenia
Evaluation of platelet response (No Response) | The time frame is up to 3 months per subject
  NR.No response (NR) was defined as platelet count < 30 × 10^9/L or a less than two fold increase in platelet count from baseline or the presence of bleeding. Platelet count must be measured on two occasions more than a day apart.

SECONDARY OUTCOMES:
Macrophage Function | two weeks
  Measure the platelet phagocytosis ability of macrophage in vitro

CONTACTS AND LOCATIONS:
Overall Officials: Jun Peng, dr., Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China